CLINICAL TRIAL: NCT01568567
Title: To Demonstrate That a Novel Powder Formulation of Lactobacillus Reuteri DSM 17938 is Safe in Adults, a Randomized, Placebo Controlled Double-blind Study
Brief Title: Study to Demonstrate the Safety of a Novel Powder Formulation of Lactobacilli in Adults
Acronym: BSSII
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Good Food Practice, Sweden (Industry)
Collaborators: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CSP U-11-008; CSUB0031 (Other Grant/Funding Number: Biogaia AB)
Record Dates: First submitted 2012-03-28; First posted 2012-04-02 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Safety
Keywords: safety; tolerance; lactobacillus Reuteri

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Double dose (Active Comparator): One stick pack with active ingredients contains 1.0 g contains 75% GOS (galactooligosaccharide), 25% L-Rhamnose, 1x108 live bacteria (CFU) Lactobacillus reuteri and silicon dioxide
  Interventions: Dietary Supplement: Lactobacillus Reuteri DSM 17938
- Single dose (Active Comparator): One stick pack with active ingredients contains 1.0 g contains 75% GOS (galactooligosaccharide), 25% L-Rhamnose, 1x108 live bacteria (CFU) Lactobacillus reuteri and silicon dioxide
  Interventions: Dietary Supplement: Lactobacillus Reuteri DSM 17938
- Placebo (Placebo Comparator): One stick pack with placebo contains 1.0 g maltodextrin and silicon dioxide
  Interventions: Dietary Supplement: Lactobacillus Reuteri DSM 17938

INTERVENTIONS:
Dietary Supplement: Lactobacillus Reuteri DSM 17938 — One stick pack in the morning and one stick pack afternoon/evening for 28 days.

SUMMARY:
Lactobacilli are commensal bacteria common to the gut of all mammals studied and traditionally associated with foods are considered safe.The established safe use on a diversity of foods and supplement products worldwide supports this conclusion. Lactobacillus reuteri is one species of Lactobacillus that naturally inhabits the gastrointestinal tract of humans and is one of the few autochthonous (indigenous) Lactobacillus species in infants as well as adults.

Although the tolerability of DSM 17938 in a tablet formulation has earlier been established, it is desirable to repeat the assessment in this novel formulation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18-65 years at visit 1
* BMI 19-29
* Hb ≥ 120 g/l for women and ≥ 130 g/l for men
* Healthy as assessed by the screening laboratory tests and blood pressure determined by the MD
* Signed informed consent and biobank consent

Exclusion Criteria:

* Participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study
* Use of oral antibiotics or probiotics during 2 weeks prior to visit 1. Other probiotics other than the study products are not allowed during the study period.
* Pregnant or lactating or wish to become pregnant during the period of the study.
* Lack of suitability for participation in the trial, for any reason, as judged by the personnel at Good Food Practice AB.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety measured by blood chemistry parameters | 28 days
  To assess the safety of a novel formulation containing Lactobacillus reuteri DSM 17938 by measuring blood chemistry parameters before and after 28 days of supplementation.
Tolerability measured by blood chemistry parameters | 28 days
  To assess tolerability of a novel formulation containing Lactobacillus reuteri DSM 17938 by measuring blood chemistry parameters before and after 28 days of supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Olsson, PhD, Principal Investigator — KPL Good Food Practice AB
Locations (1):
- Good Food Practice Uppsala, Uppsala, Sweden